CLINICAL TRIAL: NCT06969807
Title: Clinical Study to Evaluate the Efficacy and Safety of Mesenchymal Stromal Cell (Amimestrocel ) in Patients With Diabetic Kidney Disease
Brief Title: Safety and Efficacy of Mesenchymal Stromal Cells (Amimestrocel ) in Diabetic Kidney Disease
Acronym: MSC-DKD-001
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiangmei, Principal Investigator, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2025-166; S2025-166-02 (Other: Ethics Committee of Chinese PLA General Hospital)
Record Dates: First submitted 2025-04-24; First posted 2025-05-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Kidney Disease (DKD)
Keywords: mesenchymal stromal cells(MSCs); Diabetic kidney disease (DKD)
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amimestrocel (Experimental): patients receive standard treatment and Amimestrocel is administered via Intravenous infusion on day 1, 14, 28, and week 8, 12, 16, 20, 24.
  Interventions: Drug: Amimestrocel

INTERVENTIONS:
Drug: Amimestrocel — In the first month (day 1, 14, 28): 1×10E6 cells per kilogram. From the 8th to the 24th week (week 8, 12, 16, 20, 24): 1.5×10E6 cells per kilogram.

SUMMARY:
This trial is to evaluate the efficacy and safety of umbilical cord-derived mesenchymal stromal cells (Amimestrocel ) in study subjects with progressive diabetic kidney disease (DKD), to investigate whether Amimestrocel can improve renal function or proteinuria of DKD patients.

ELIGIBILITY:
Inclusion Criteria: -

1. Men and women who are ≥ 45 and ≤ 80 years old.
2. Diagnosed with type 2 diabetes mellitus.
3. Diagnosed with diabetic kidney disease based on renal pathology within the past 10 years.
4. The 24-hour urine protein quantification is continuously ≥ 3.5 g, and the urine albumin-to-creatinine ratio (UACR) > 1000 mg/g.
5. The estimated glomerular filtration rate (eGFR) ≥ 20 ml/min/1.73m² (calculated according to the CKD-EPI formula).
6. The blood pressure can be controlled at BP ≤ 160/100 mmHg.
7. Glycated hemoglobin (HbA1c) < 9%.
8. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Patients with kidney diseases not caused by diabetes mellitus.
2. Patients who have received treatment with systemic immunosuppressants (such as cyclosporine A, tacrolimus, mycophenolate mofetil, etc.) within 30 days before enrollment and the duration of treatment exceeds one week.
3. Severe cardiovascular diseases, such as congenital heart diseases, atrial fibrillation, NYHA class Ⅲ-IV, unstable angina pectoris, etc.
4. A history of cerebral hemorrhage or cerebral infarction within the past six months (except for those with a history of lacunar cerebral infarction without residual limb movement disorders, cognitive and language function disorders).
5. Patients with severe hyperlipidemia: (serum triglyceride ≥ 6.2 mmol/L, serum low-density lipoprotein cholesterol ≥ 4.1 mmol/L).
6. Hyperkalemia that cannot be controlled through diet or potassium-lowering treatment.
7. Patients with active infections of hepatitis B or hepatitis C viruses (the copy number of HBV DNA or HCV RNA exceeds the upper limit of the normal value); patients with active tuberculosis; patients with severe immunodeficiency diseases, human immunodeficiency virus (HIV) infection, etc.
8. Patients with a history of malignant tumors within the past five years.
9. Patients with a known history of severe allergy to component blood or blood products, or patients with a history of allergy to heterologous proteins.
10. Lactating women, or female patients who have a pregnancy plan or an egg donation plan from the start of the study to the follow-up period, and male patients (or their partners) who have a childbearing plan or a sperm donation plan from the start of the study to the follow-up period and are unwilling to take contraceptive measures.
11. Active infection within one week before enrollment and requiring treatment with intravenous antibiotics.
12. Patients who have participated in other interventional clinical trials within three months before enrollment.
13. The research physician deems that the patient's condition is not suitable for participating in this clinical study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Urine protein | Change from baseline at 28 weeks
  Urine protein will be measured on 24h urine samples
estimated Glomerular Filtration Rate(eGFR) | Change from baseline at 28 weeks
  GFR will be estimated by CKD-EPI

SECONDARY OUTCOMES:
fasting blood glucose | Change from baseline at 28 weeks and then every 6 months to study completion, up to 24 months after cell infusion
  fasting blood glucose
HbA1c | Change from baseline at 28 weeks and then every 6 months to study completion, up to 24 months after cell infusion
  Glycated Hemoglobin A1c
Urinary Albumin/Creatinine Ratio(UACR) | Change from baseline at 28 weeks and then every 6 months to study completion, up to 24 months after cell infusion
  UACR will be measured on spot morning urine samples
proportion of outcome ( ≥50% declined in eGFR，reached end stage renal disease (ESRD), or occured Renal replacement) | proportion of study participants within outcome at 28 weeks and then every 6 months to study completion, up to 24 months after cell infusion
  proportion of outcome ( ≥50% declined in eGFR，reached End Stage Renal Disease (ESRD), or occured Renal Replacement Therapy)
proportion of major adverse cardiac events(MACE) and all-cause mortality | proportion of study participants within outcome at 28 weeks and then every 6 months to study completion, up to 24 months after cell infusion
  proportion of major adverse cardiac events(MACE:CV death, non-fatal CV event(myocardial infarction, stroke, hospitalization for HF)) and all-cause mortality
Mechanism exploration | Change from baseline at 4,12,28 weeks and 12 months
  Explore the mechanism through blood tests（Serum/plasma concentrations (pg/ml) of biomarkers of inflammation. Proportion/total number of circulating T cells, B cells, NK cells, etc ）.
changes in retinal imaging | Change from baseline at 28 weeks and then every 6 months to study completion, up to 24 months after cell infusion
  Macular vascular density by Optical Coherence Tomography Angiography （OCTA）， and analyze the percentage of changes in retinal imaging of patients compared to the baseline .
Changes in peripheral nerve injury | Change from baseline at 28 weeks and then every 6 months to study completion, up to 24 months after cell infusion
  Examine through electromyography, to evaluate the percentage of changes in peripheral nerve injury of patients compared with the baseline.
Changes in symptoms | Change from baseline at 28 weeks and then every 6 months to study completion, up to 24 months after cell infusion
  The traditional Chinese Medicine（TCM）Syndrome Rating Scale will be used to score TCM symptoms，to evaluate the percentage of changes in the symptoms of patients compared with the baseline.
Changes in the quality of life scale | Change from baseline at 28 weeks and then every 6 months to study completion, up to 24 months after cell infusion
  The Diabetes Quality-of-Life Measure (DQOL) will be used to score quality of life at each visit, to evaluate the percentage of the change in the DQOL of patients compared to the baseline
Adverse Event and Serious Adverse Event（SAE） | within 28 weeks after received Amimestrocel
secondary malignant disease | within 24 months after received Amimestrocel
  Number of Participants with secondary malignant disease

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Medical Center, Tsinghua University, Beijing, Beijing Municipality